CLINICAL TRIAL: NCT02333162
Title: A Phase I Study of Intensity Modulated Total Marrow Irradiation (IMTMI) in Addition to Fludarabine/Melphalan Conditioning for Allogeneic Transplantation for Advanced Hematologic Malignancies
Brief Title: Intensity Modulated Total Marrow Irradiation, Fludarabine Phosphate, and Melphalan in Treating Patients With Relapsed Hematologic Cancers Undergoing a Second Donor Stem Cell Transplant
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-0709; NCI-2014-02469 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB14-0709 (Other: University of Chicago Comprehensive Cancer Center); P30CA014599 (NIH)
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Previously Treated Myelodysplastic Syndrome; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Hematologic Malignancy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Hematologic Neoplasms | interventions — fludarabine phosphate; Melphalan; Radiotherapy, Intensity-Modulated; Peripheral Blood Stem Cell Transplantation; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (IMTMI, combination chemotherapy, PBSCT or BMT) (Experimental): CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 30 minutes daily on days -7 to -3 and melphalan IV on day -2. Patients also undergo IMTMI BID for 2 to 5 days between days -7 to -3.
  TRANSPLANT: Patients undergo allogeneic PBSCT or BMT on day 0.
  GVHD PROPHYLAXIS: Patients receive tacrolimus IV continuously over 24 hours or PO BID on days -2 to 180 with taper thereafter and mycophenolate mofetil IV every 8 hours or PO on days 0-28 (for matched donors) or days 0-40 (for alternative donors) with taper to day 60.
  Interventions: Drug: Fludarabine Phosphate; Drug: Melphalan; Radiation: Intensity-Modulated Radiation Therapy; Radiation: Total Marrow Irradiation; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Procedure: Allogeneic Bone Marrow Transplantation; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; SH T 586
Drug: Melphalan — Given IV
  Other Names: Alkeran
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMTMI
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Radiation: Total Marrow Irradiation — Undergo IMTMI
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic PBSCT
  Other Names: HSC; HSCT
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic PBSCT
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Procedure: Allogeneic Bone Marrow Transplantation — Undergo allogeneic BMT
  Other Names: Allo BMT; Allogeneic BMT
Drug: Tacrolimus — Given IV or PO
  Other Names: Advagraf; FK 506
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: Cellcept; MMF
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and the best dose of intensity modulated total marrow irradiation (IMTMI) when given together with fludarabine phosphate and melphalan in treating patients with cancers of the blood (hematologic) that have returned after a period of improvement (relapsed) undergoing a second donor stem cell transplant. IMTMI is a type of radiation therapy to the bone marrow that may be less toxic and may also reduce the chances of cancer to return. Giving fludarabine phosphate, melphalan, and IMTMI before a donor stem cell transplant may help stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The determine the maximum tolerated dose (MTD) of intensity-modulate total marrow irradiation (IMTMI) in combination with fludarabine (fludarabine phosphate)/melphalan as conditioning for second allogeneic stem cell transplantation for patients with hematologic malignancies.

SECONDARY OBJECTIVES:

I. To determine the overall toxicity and day 100 transplant related mortality after second allogeneic hematopoietic stem cell transplantation conditioned with increasing doses of intensity-modulate total marrow irradiation (IMTMI) in combination with fludarabine/melphalan.

II. To determine the time to neutrophil and platelet engraftment after second allogeneic hematopoietic stem cell transplantation conditioned with increasing doses of intensity-modulate total marrow irradiation (IMTMI) in combination with fludarabine/melphalan.

III. To determine the overall survival (OS) and event-free-survival (EFS) in patients with hematologic undergoing second allogeneic hematopoietic stem cell transplant (HSCT) after conditioning with fludarabine/melphalan and IMTMI.

OUTLINE: This is a dose-escalation study of IMTMI.

CONDITIONING REGIMEN: Patients receive fludarabine phosphate intravenously (IV) over 30 minutes daily on days -7 to -3 and melphalan IV on day -2. Patients also undergo IMTMI twice daily (BID) for 2 to 5 days between days -7 to -3.

TRANSPLANT: Patients undergo allogeneic peripheral blood stem cell transplant (PBSCT) or bone marrow transplant (BMT) on day 0.

GRAFT-VERSUS-HOST DISEASE (GVHD) PROPHYLAXIS: Patients receive tacrolimus IV continuously over 24 hours or orally (PO) BID on days -2 to 180 with taper thereafter and mycophenolate mofetil IV every 8 hours or PO on days 0-28 (for matched donors) or days 0-40 (for alternative donors) with taper to day 60.

After completion of treatment, patients are followed up periodically for 1 year and then yearly for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following diseases: acute myeloid leukemia (AML) and high risk myelodysplastic syndrome (MDS) undergoing second allogeneic (allo)-stem cell transplant (SCT) using the same donor or different donor for disease relapse; patients with other hematologic malignancies, including acute lymphoblastic leukemia (ALL), will be at the discretion of the investigators
* Karnofsky performance status of 70 or above
* Life expectancy is not severely limited by concomitant illness
* Adequate cardiac and pulmonary function; patients with decreased left ventricular ejection fraction (LVEF) =< 40% or diffusion capacity of carbon monoxide (DLCO) =< 50% of predicted will be evaluated by cardiology or pulmonary prior to enrollment on this protocol
* Serum creatinine =<1.5 mg/dL or creatinine clearance > 50 ml/min; some patients with minor deviations may be accepted on protocol after discussion with the principal investigator (PI)
* Serum bilirubin =< 2.0 mg/dl; some patients with minor deviations may be accepted on protocol after discussion with the PI
* Serum glutamic oxaloacetic transaminase (SGPT) < 5 x upper limit of normal; some patients with minor deviations may be accepted on protocol after discussion with the PI
* No evidence of chronic active hepatitis or cirrhosis
* Human immunodeficiency virus (HIV)-negative
* Patient is not pregnant
* Patient or guardian able to sign informed consent
* DONOR: Since these patients already had first allo-SCT; in the majority time, the same matched donor has been used for second allo-SCT; if the patients have multiple donors, alternative matched (8/8 or 10/10) donor could be used for the second allo-SCT; the donor could be matched related donors or matched unrelated donors from registry
* DONOR: If more than one potential volunteer unrelated donor is considered suitable, further selection of the most suitable donor will be prioritized as follows or will follow our institutional guideline from our stem cell transplant standard operating procedure (SOP):

  * Age of donor (18-24 > 25-34 > 35-44 > 45+)
  * Sex of donor (male > female, nulliparous female > parous, multiparous female)
  * Cytomegalovirus (CMV) status, if recipient is CMV seronegative (CMV- > CMV+

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-12-05 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
MTD of conditioning regimen defined as any grade III or higher dose-limiting toxicity, graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 30 days post second allo-SCT

SECONDARY OUTCOMES:
Overall incidence of adverse events, graded according to the NCI CTCAE version 4.0 | Up to 2 years
Transplant related mortality | Day 100
Time to neutrophil engraftment | First day in which the ANC is > 500/mm^3 for 3 consecutive days
Time to platelet engraftment | First day the platelet count is > 20,000/mm^3 without transfusion support for 7 consecutive days
overall survival (OS) | Up to 2 years
event-free-survival (EFS) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hongtao Liu, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States